CLINICAL TRIAL: NCT05660707
Title: Patients Who Underwent Surgical Procedures State of Readiness for Discharge: Mixed Methods Research
Brief Title: Patients Who Underwent Surgical Procedures State of Readiness for Discharge
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma CEBECİ, Principal Investigator, Akdeniz University
Other Study IDs: KAEK-959-2021
Record Dates: First submitted 2022-12-09; First posted 2022-12-21 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2022-12

CONDITIONS: Surgery; Patients; Discharge Readiness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, it was aimed to evaluate the readiness status of patients who are planned to be discharged after the surgical procedure.

DETAILED DESCRIPTION:
Objective: In this study, it was aimed to evaluate the readiness status of patients who are planned to be discharged after the surgical procedure.

Method: Explanatory sequential mixed design will be used in accordance with the purpose of the study. The purpose of the exploratory sequential design is to clarify the relationships obtained with the quantitative data by applying the qualitative step.

This pattern is applied in two stages. The first phase begins with the collection of quantitative data that will essentially answer the research question. In the second stage, qualitative data are collected and the collected data is interpreted to help explain the quantitative results.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Willingness and willingness to participate in the study,
* Having undergone a surgical procedure,
* Healing / discharge as it is,
* Not having difficulties in understanding
* Patients who do not feel ready for discharge according to quantitative data and also agree to participate in the qualitative study

Exclusion Criteria:

* Be under the age of 18,
* Being discharged without surgical procedure,
* Transfer to another department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the Turkish validity and reliability study, the minimum sample size for the 95% confidence interval was calculated as 1251 (t=1.96; d=0.1) by using the standard deviation value (σ=1.85) found for the Discharge Readiness Scale.
  Considering that there would be missing or missing data, it was planned to take 10% more than the number of samples.
  As a result, the number of samples was determined as 1376.
Sampling Method: Non-Probability Sample
Enrollment: 870 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Readiness status of patients whose discharge is planned | within 24 hours before discharge
  Readiness for Hospital Discharge Scale/Short Form

SECONDARY OUTCOMES:
Reasons why patients are not ready for discharge | within 24 hours before discharge
  semi-structured interview form

CONTACTS AND LOCATIONS:
Overall Officials: Fatma CEBECİ, Prof., Principal Investigator — Akdeniz University; Songül BİŞKİN ÇETİN, PhD., Study Chair — Akdeniz University; Arzu TAT ÇATAL, RN, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)